CLINICAL TRIAL: NCT00006499
Title: Genetics of Hypertension and Its Intermediate Phenotypes
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 940; R01HL064109 (NIH)
Record Dates: First submitted 2000-11-16; First posted 2000-11-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-07

CONDITIONS: Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

SUMMARY:
To define the underlying genetics of hypertension in an Asian population by studying intermediate phenotypes.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension, an exceedingly common trait in most developed countries, imparts an increased risk of cardiovascular, cerebrovascular and renal diseases. Nevertheless, the primary determinants of elevated blood pressure in most patients are unknown. Recognizing that a sizable portion of variation in blood pressure is genetically determined, one line of research has focused on identifying genetic variants that contribute to the pathogenesis of hypertension. However, standard genetic linkage analysis using "hypertension" as a phenotype may lack power due to the multifactorial nature of the disorder. A way to overcome this challenge is to subdivide hypertensive subjects into more homogenous subgroups.

DESIGN NARRATIVE:

The overall goal, which is to define the underlying genetics of hypertension in an Asian population by studying intermediate phenotypes, can be divided into three parts. First, the rural Chinese population will be characterized by the collection of intermediate phenotype data on 600 unrelated individuals with high diastolic blood pressure and on 100 normotensive controls. Intermediate phenotypes include: 1) non-modulation of adrenal and renal vascular responses to angiotensin II with changes in sodium intake; 2) altered urinary kallikrein excretion; 3) low plasma renin activity response to volume depletion; 4) increased free cortisol excretion; and 5) insulin resistance. Second, candidate genes will be chosen according to the underlying physiology of the intermediate phenotypes, and variations in the coding sequences of these potentially relevant genes will be identified. Finally, polymorphisms identified in the candidate genes will be tested through case-control analyses defined by the intermediate phenotypes.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-06; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiping Xu — Harvard University School of Public Health